CLINICAL TRIAL: NCT04128618
Title: A Randomized, Sham Controlled, Double-blind, Multi-center Study of Neuromuscular Electrical Stimulation (NMES) as an Adjunctive Therapy for Knee Pain Relief and Improving Functional Outcomes in Knee Osteoarthritis (OA) Patients
Brief Title: Evaluation of a Home-based NMES Therapy for Knee Osteoarthritis Pain
Acronym: NMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CyMedica Orthopedics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CM-2019
Record Dates: First submitted 2019-10-07; First posted 2019-10-16 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Knee Osteoarthritis
Keywords: knee OA; arthritis; knee pain
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects, coordinators, and Investigators are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active NMES (Experimental)
  Interventions: Device: CyMedica e-vive NMES
- Modified NMES sham (Sham Comparator)
  Interventions: Device: CyMedica e-vive NMES

INTERVENTIONS:
Device: CyMedica e-vive NMES — Neuromuscular Electrical Stimulation (NMES) therapy

SUMMARY:
Evaluation of knee pain and functional mobility of knee osteoarthritis patients with a home-based neuromuscular electrical stimulation (NMES) therapy

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written, informed consent before any study procedures occur. The subject should be provided with a copy of the signed Informed Consent upon signature.
2. Subjects with symptomatic Kellgren-Lawrence (KL) Grade 2, 3, or 4 OA by radiograph (AP tunnel view) within 30 days prior to day 0 visit, where the K-L grades are defined as:

   * Grade 0: no radiographic features of OA are present
   * Grade 1: doubtful joint space narrowing (JSN) and possible osteophytic lipping
   * Grade 2: definite osteophytes and possible JSN on anteroposterior weight-bearing radiograph
   * Grade 3: multiple osteophytes, definite JSN, sclerosis, possible bony deformity
   * Grade 4: large osteophytes, marked JSN, severe sclerosis and definite bony deformity
3. Subject must have a normal tibiofemoral angle (0-8°) and a joint space width of ≥ 3mm confirmed by radiograph.
4. Subjects who are between the ages of 21 - 85 years.
5. Subjects must have a visual analog pain (VAS) score of at least 4 cm on a 10 cm scale for a nominated activity in the target knee at the time of screening.
6. For bilateral knee osteoarthritis subjects, the visual analog pain VAS score for a nominated activity of the contralateral knee must be less than 4 cm on the VAS scale.
7. Subject has access to a smartphone or tablet (Android or iOS).
8. Subject must be ambulatory.
9. Subject must be willing to discontinue receiving knee intra-articular injections of steroids, knee intra-articular injections of hyaluronic acid, opioids, and analgesics (except for acetaminophen up to 3000 mg/day or an equivalent) for the duration of the study.
10. Subject must be willing to take acetaminophen (up to 3000 mg/day) or an equivalent as pain medication for the duration of the study.
11. Subject must be willing to stop taking any pain medications 24 hours prior any scheduled study visit.
12. Subject must be willing to stop receiving knee physical therapy of the target knee for the duration of the study.
13. Subject must be willing to stop wearing any knee unloader brace of the target knee for the duration of the study.
14. Subjects must be proficient in English.
15. Subjects must be willing and able to comply with all study procedures for the duration of the clinical study

Exclusion Criteria:

1. Subjects who have a body mass index ≥ 40 at the time of consent (at the discretion of the PI).
2. Subjects with a diagnosis of inflammatory arthritis (knee rheumatoid arthritis, active gout, knee joint infection, Lyme disease, SLE, etc.).
3. Subjects with a diagnosis of severe neuropathy condition for the past 6 months and under medication for treatment of the condition.
4. Subjects with a diagnosis of fibromyalgia for the past year.
5. Subjects who have had an injury or an acute traumatic injury to the target knee within 6 months of screening.
6. Subject must NOT have had arthroscopy of the target knee within 8 weeks of randomization.
7. Subjects who have had treatment of the target knee with intra-articular injections of steroids within 8 weeks of screening.
8. Subjects who have had intra-articular injections of hyaluronic acid within 12 weeks of screening.
9. Subjects who have had a scheduled surgery on the target knee within the study period.

   (Note- Subjects who are scheduled to go under total knee replacement surgery within the next 3 months at screening will not be enrolled. Subjects that are contemplating the surgery can be included.)
10. Subjects who have used electrotherapy or acupuncture for OA of the target knee within 4 weeks of screening.
11. Subjects who have used Neuromuscular Electrical Stimulation (NMES) in the past year.
12. Subjects with significant and clinically evident mal-alignment of the target knee (> 5 degrees varus or valgus in the target knee).
13. Subjects with surgical metallic hardware in the target knee.
14. Subjects who have had implanted electrical devices (cardiac pacemakers, deep brain stimulators, implantable cardiac defibrillators).
15. Subjects who have contraindications to X-rays.
16. Subjects with a current malignancy or who have received treatment for malignancy with the last 5 years, with the exception of resected basal cell carcinoma and squamous cell carcinoma of the skin.
17. Subjects who have an active substance abuse problem (drugs or alcohol) or a history of chronic substance abuse (> 5 years).
18. Subjects with skin breakdown or infection in the area where the study device will be placed (quadriceps of the target knee).
19. Subjects with any chronic conditions (e.g., diabetes, hypertension, congestive heart failure, etc.) that have not been well-controlled for at least 3 months prior to screening.
20. Subjects who have any ongoing litigation for worker's compensation.
21. Subjects with any condition, in the opinion of the Investigator that might interfere with the evaluation of the study objectives.
22. Subjects who are pregnant.
23. Subject must not have participated in a clinical study within the past 12 weeks from the last day of treatment that required the use of an investigational device, drug or biologic

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Knee pain using VAS scale (Visual Analog Scale) | 12 weeks post intervention
  Pain associated with knee osteoarthritis- Unit none (score)

SECONDARY OUTCOMES:
Timed Up & Go (TUG) | 12 weeks post intervention
  Mobility and functionality assessment of the knee- Timed Up & Go (TUG), unit seconds
Quadriceps muscle strength | 12 weeks post intervention
  Strength assessment, Quadriceps strength using a handheld dynamometer, unit lbs/in
Repeated Chair Rise | 12 weeks post intervention
  Mobility and functionality assessment of the knee- Repeated chair rise, unit none (number of times)
3 min walk test | 12 weeks post intervention
  Mobility and functionality assessment of the knee- 3 min walk test, unit meters
KOOS JR. Survey | 12 weeks post intervention
  Mobility and functionality assessment of the knee- KOOR JR- Unit, none (score)
WOMAC Survey | 12 weeks post intervention
  Mobility and functionality assessment of the knee- WOMAC- Unit, none (score)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Noble Clinical Research, Tucson, Arizona
  - Site 1, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No